CLINICAL TRIAL: NCT02124122
Title: Safety of Lactobacillus Reuteri in Healthy Children Ages 2 to 5 Years in Peru
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tulane University School of Medicine (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH); Johns Hopkins Bloomberg School of Public Health (Other); Asociacion Benefica Prisma (Other)
Responsible Party: Principal Investigator, Richard A. Oberhelman, Professor, Tulane University School of Medicine
Organization: Tulane University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FDA IND# 13710-Protocol 2; 5U01AT002733 (NIH)
Record Dates: First submitted 2014-04-24; First posted 2014-04-28 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: Focus; safety

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lactobacillus (Experimental): Lactobacillus reuteri (Lr): 108 (100 million) organisms of Lactobacillus reuteri per dose, given once daily for a five-day treatment period that corresponds to a dose of the closely related L. reuteri ATCC 55730 strain that has shown to be therapeutic for infantile colic. The strain used in this study (DSM 17938) has been cured of an antibiotic resistance plasmid found in the original BioGaia strain (L. reuteri ATCC 55730).
  Interventions: Biological: Lactobacillus reuteri
- Placebo (Placebo Comparator): Placebo oil preparation, administered as 5 drops of the oil vehicle used in manufacturing the Lr suspension, given once daily for a five-day study period (BioGaia AB, Stockholm, Sweden).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Lactobacillus reuteri — Probiotic
  Other Names: BioGaia Probiotic Drops
  Arms: Lactobacillus
Biological: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a Phase 1 study to assess the safety and tolerability of Lactobacillus reuteri (Lr) strain DSM 17938 in healthy children in Peru. It is a preliminary study in support of a clinical trial to assess safety and efficacy of L. reuteri for treatment of pediatric diarrhea in Peru.

DETAILED DESCRIPTION:
This is a phase I blinded randomized study of the safety and tolerability of Lactobacillus reuteri DSM 17938 given daily for a period of five consecutive days. Upon enrollment subjects will be randomized to one of two treatment groups in a ratio of treatment to placebo of 2:1. Subjects will be randomized to receive either:

A. Lactobacillus reuteri (Lr): 108 (100 million) organisms of Lactobacillus reuteri per dose, given once daily for a five-day treatment period that corresponds to a dose of the closely related L. reuteri ATCC 55730 strain that has shown to be therapeutic for infantile colic. The strain used in this study (DSM 17938) has been cured of an antibiotic resistance plasmid found in the original BioGaia strain (L. reuteri ATCC 55730).

B. Placebo oil preparation, administered as 5 drops of the oil vehicle used in manufacturing the Lr suspension, given once daily for a five-day study period (BioGaia AB, Stockholm, Sweden).

In the first 30 subjects randomized, administration of each dose of the study preparation drops (A or B above) will be immediately followed by offering 2 ounces of flavored PediaSure ® (Abbott Laboratories) nutritional supplement to each child. The second 30 subjects enrolled will not be offered PediaSure ® after product administration. This format will also allow us to assess the impact of concurrent administration of a buffering non-lactose containing formula with prebiotic nutritional properties on intestinal colonization with L. reuteri by PCR.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 2-5 years with no exclusion criteria

Exclusion Criteria:

* 1) No enrollment of family members in households where any of the following are present:

  1. Another study participant in the household
  2. Pregnancy or current breastfeeding by any household member
  3. Presence of an infant under age 6 months living in the household
  4. Presence of immune suppressed individuals or use of immunosuppressive agents (including but not limited to corticosteroids and methotrexate, etc.) by any household member
  5. Presence of a serious congenital anomaly or chronic medical condition that in the opinion of the investigators would contraindicate participation in any household member, including history of gastrointestinal surgery, chronic gastrointestinal illness, abnormal intestinal anatomy, or abnormal bowel functionality

     2) Allergy to penicillin or cephalosporins or gentamicin 3) History of antibiotic use in the last 30 days 4) Use of probiotic products within the past 90 days, including masato (local product with fermenting bacteria) and yogurt products containing live bacterial cultures.

     5) History of diarrheal illness within the past 30 days 6) Presence of fever or a pre-existing adverse event monitored in the study 7) Positive results on serum diagnostic tests for antibodies to HIV.

     Testing for Hepatitis B core antigen, and Hepatitis C is not necessary in children as in adults, since there is universal vaccination for Hepatitis B among children in this community, and both forms of hepatitis are rare and largely asymptomatic in this age group.

     8) Presence of severe anemia, defined as serum hemoglobin < 8 gm/dL

     9) Out of range laboratory values for tests monitored as potential adverse events, as described in Appendix 2, B. LABORATORY VALUES, and detected based on Day 0 blood test results. However, subjects will only be excluded based on serum hemoglobin if they meet exclusion criterion 8.

     10) Pre-enrollment stool sample (collected within 14 days of Day 1 of the study) is positive for L. reuteri by PCR.

Ages: 2 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2015-03; Primary Completion 2015-11 (Actual); Study Completion 2016-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard A Oberhelman, MD, Principal Investigator — Tulane School of Public Health and Tropical Medicine; Margaret N Kosek, MD, Study Director — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Community of Santa Clara, Santa Clara, Loreto, Peru

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kosek MN, Penataro-Yori P, Paredes-Olortegui M, Lefante J, Ramal-Asayag C, Zamora-Babilonia M, Meza-Sanchez G, Oberhelman RA. Safety of Lactobacillus Reuteri DSM 17938 in Healthy Children 2-5 Years of Age. Pediatr Infect Dis J. 2019 Aug;38(8):e178-e180. doi: 10.1097/INF.0000000000002267. PMID 30531312

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Lactobacillus | Placebo
Started | 41 | 19
Completed | 41 | 19
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Lactobacillus | Placebo | Total
Number analyzed (Participants) | 41 | 19 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 4.04 (1.278) | 3.31 (1.080) | 3.81 (1.258)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 13 | 34
  Male | 20 | 6 | 26
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 41 | 19 | 60
  Not Hispanic or Latino | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Peru | 41 | 19 | 60

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Positive Blood Culture for L Reuteri
Time Frame: Participants are followed an average of 36 days
Measure: Count of Participants; unit: Participants
Arm/Group | Lactobacillus | Placebo
Number analyzed (Participants) | 41 | 19
Participants | 0 | 0

2. Primary Outcome: Mean Daily Temperature
Description: Mean of body temperatures recorded on study days listed, averaged across all participants at all time points
Time Frame: Study days 1-5, 8,12, 15, 18, 28, and 36
Measure: Mean (Standard Deviation); unit: Degrees Celsius
Arm/Group | Lactobacillus | Placebo
Number analyzed (Participants) | 41 | 19
Degrees Celsius | 36.50 (0.288) | 36.45 (0.232)

ADVERSE EVENTS:
Time Frame: Day 0 through Day 28 after day 0
Arm/Group | Lactobacillus | Placebo
Serious Adverse Events (participants affected / at risk) | 0/41 | 0/19
Other Adverse Events (participants affected / at risk) | 25/41 | 18/19
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Lactobacillus (N=41) | Placebo (N=19)
Diarrhea (Gastrointestinal disorders) | 4 (6) | 7 (7) — At least one episode of diarrhea during 28 days of active surveillance
Upper repiratory infection (Respiratory, thoracic and mediastinal disorders) | 23 (32) | 9 (14)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Urinary tract infection (Renal and urinary disorders) | 3 (3) | 2 (2)
Cellulitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 1 (1)
Scabies (Infections and infestations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No